CLINICAL TRIAL: NCT03145519
Title: A Randomized Controlled Trial to Demonstrate the Safety and Efficacy of the OptiVein IV Catheter In a Pediatric Population
Brief Title: A Trial to Demonstrate the Safety and Efficacy of the OptiVein IV Catheter In a Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optomeditech Oy (Industry)
Collaborators: CardioMed Device Consultants, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMT-CT-004-PED
Record Dates: First submitted 2017-02-20; First posted 2017-05-09 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Injections, Intravenous; Administration, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OptiVein (Experimental): Placement of IV-catheter and administration of treatment using OptiVein catheter.
  Interventions: Device: OptiVein Catheter
- Vasofix Certo (Active Comparator): Placement of IV-catheter and administration of treatment using Vasofix Certo catheter.
  Interventions: Device: Vasofix Certo Catheter

INTERVENTIONS:
Device: Vasofix Certo Catheter — Placement of IV-catheter
  Arms: Vasofix Certo
Device: OptiVein Catheter — Placement of IV-catheter
  Arms: OptiVein

SUMMARY:
A prospective, single-center, open-label, randomized controlled trial to demonstrate the safety and efficacy of the OptiVein IV Catheter in the pediatric population. The study hypothesis is that OptiVein IV Catheter use will be superior to the control in successful venous access after first attempt.

DETAILED DESCRIPTION:
The OptiVein IV Catheter is a sterile single use disposable intravascular cannulation device that is modified from CE certified Vasofix Certo Catheter from B.Braun with the additional features of an optical fiber and modified flashplug. The OptiVein System also includes an electronic unit.

The OptiVein Catheter shares a similar intended use and the same catheter components as the Vasofix Certo IV Catheter. Clinical data will be obtained to demonstrate that there is no change to the safety and efficacy profile due to the laser component of the OptiVein IV Catheter.

A prospective, single-center, open-label, randomized controlled trial to demonstrate the safety and efficacy of the OptiVein IV Catheter in the pediatric population. The study hypothesis is that OptiVein IV Catheter use will be superior to the control in successful venous access after first attempt.

Patients aged newborn to twelve (12) years requiring short-term use of an IV catheter to withdraw blood samples or to administer fluids or medications intravenously.

Participating sites will follow routine practice guidelines regarding the personnel responsible for inserting the catheters for this study, known herein as "operators." Operators must be professionally trained in IV catheter placement; educational background and level of experience of operator will be documented.

All Operators selected for participation in the study will undergo training on the protocol, Good Clinical Practice and the assembly and use of the OptiVein IV Catheter and Vasofix Certo IV catheter prior to enrolling patients into the study.

Randomization will be in a 1:1 fashion with assignment given by the electronic data capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

* Aged newborn to 12 years
* Has written or verbal order for insertion of an IV
* Requires peripheral IV therapy (catheter)
* Has an insertion site in the forearm, hand, foot, leg, or head free of deformities, phlebitis, infiltration, dermatitis, burns, lesions or tattoos
* Demonstrates cooperation with a catheter insertion and the study protocol
* Informed consent has been obtained

Exclusion Criteria:

* Life expectancy less than 72h.
* Any child the research staff deem unobservable
* The study IV catheter site will be placed below an old infusion site
* Will likely require a power injection for a radiologic procedure during participation in this study

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | Immediate / During the procedure usually taking less than 1 minute
  Successful IV insertion on the first attempt, defined as placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.

SECONDARY OUTCOMES:
Number of attempts | Immediate / During the consecutive attempts to place the catheter, usually less than 30 minutes
  Total number of attempts required for successful IV insertion.
Time to successful IV insertion | Immediate / During the procedure usually taking less than 1 minute if successful with first stick or within 30 minutes if further attempts are required
  Time to successful IV insertion, defined as time from the first skin puncture to placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal
Incidence of blood extravasation resulting in a hematoma | Immediate / 72 hour follow-up or time of removal of catheter, whichever occurs first
Incidence of fluid extravasation delivered through catheter | Immediate / 72 hour follow-up or time of removal of catheter, whichever occurs first
Incidence of infection | 72 hour follow-up or time of removal of catheter, whichever occurs first
  Incidence of infection (phlebitis, dermatitis and induration) at insertion site through 72 hours or at the time of catheter removal, whichever occurs first.
Unplanned withdrawal of IV catheter | 72 hour follow-up or time of removal of catheter, whichever occurs first
Overall complication rate composed from #2-5 above | 72 hour follow-up or time of removal of catheter, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Tuuli Metsvaht, MD, Principal Investigator — Tartu University Hospital, Children's Clinic
Locations (1):
- Tartu University Hospital, Children's Clinic, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No